CLINICAL TRIAL: NCT04857138
Title: An Open-Label, Multicenter, Dose-Escalation and Expansion, Phase I Study to Evaluate Safety, Pharmacokinetics, And Anti-Tumor Activity of RO7300490, A Fibroblast Activation Protein-α (FAP) Targeted CD40 Agonist, as Single Agent or in Combination With Atezolizumab in Participants With Advanced and/or Metastatic Solid Tumors
Brief Title: A Study to Evaluate Safety, Pharmacokinetics and Anti-Tumor Activity of RO7300490, as Single Agent or in Combination With Atezolizumab in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WP42627; 2020-004489-21 (EudraCT Number)
Record Dates: First submitted 2021-04-22; First posted 2021-04-23 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose Escalation (RO7300490 Monotherapy) (Experimental): Participants will receive escalating doses of RO7300490 intravenously (IV) as a single agent for up to 24 months maximum or until progressive disease, unacceptable toxicities, death, or withdrawal of consent.
  Interventions: Drug: RO7300490
- Part 2: Dose Escalation (RO7300490/atezolizumab combination therapy) (Experimental): Participants will receive escalating doses of RO7300490 in combination with a fixed dose of atezolizumab IV (as per label) for up to 24 months maximum or until progressive disease, unacceptable toxicities, death, or withdrawal of consent.
  Interventions: Drug: RO7300490; Drug: Atezolizumab
- Part 3: Dose Expansion (Disease-specific Expansion(s)) (Experimental): Participants with selected types of advanced and/or metastatic tumors will receive the maximum tolerated dose (MTD) or recommended dose for expansion (RDE) (determined from Parts 1 and 2) of RO7300490 in combination with a fixed dose of atezolizumab IV (as per label). Treatment will be administered for up to 24 months maximum or until progressive disease, unacceptable toxicities, death, or withdrawal of consent.
  Interventions: Drug: RO7300490; Drug: Atezolizumab

INTERVENTIONS:
Drug: RO7300490 — Participants will receive RO7300490, as described in the Arm Descriptions.
Drug: Atezolizumab — Participants will receive Atezolizumab, as described in the Arm Descriptions.
  Arms: Part 2: Dose Escalation (RO7300490/atezolizumab combination therapy); Part 3: Dose Expansion (Disease-specific Expansion(s))

SUMMARY:
A study to evaluate the safety, pharmacokinetics and anti-tumor activity of RO7300490 as a single agent or in combination with atezolizumab. The study will consist of 3 parts: [Part 1] Dose-Escalation of RO7300490 as a single agent; [Part 2] Dose-Escalation of RO7300490 in combination with atezolizumab and [Part 3] Dose-Expansion of RO7300490 in combination with atezolizumab in selected cancer types.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of >= 12 weeks.
* Histologically confirmed diagnosis of locally advanced and/or metastatic solid tumors that are not amenable to standard therapy.
* Radiologically measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Agreement to provide protocol-specific biopsy material.
* Adverse Events (AEs) from prior anti-cancer therapy resolved to Grade =<1.
* Adequate performance status and cardiovascular, hematological, liver, renal and coagulation function.
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse), use contraceptive measures and refrain from donating eggs.
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse), use contraceptive measures and refrain from donating sperm.

Exclusion Criteria:

* Known central nervous system (CNS) primary tumors or metastases, including leptomeningeal metastases, unless protocol-specific conditions are met.
* Active second invasive malignancy within two years prior to screening.
* Significant cardiovascular/cerebrovascular disease within 6 months prior to study treatment start.
* Any other diseases, metabolic dysfunction, physical examination finding or clinical laboratory finding that gives reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug.
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
* Active or history of autoimmune disease.
* Known hypersensitivity to any of the components of RO7300490 formulation or to components of atezolizumab formulation.
* Pregnancy, lactation or breastfeeding.
* Dementia or altered mental status that would prohibit informed consent.
* Major surgery or significant traumatic injury within 28 days prior to the first study drug administration (excluding biopsies) or anticipation of the need for major surgery during study treatment.
* Treatment with radiotherapy, chemotherapy, hormonal therapy, targeted therapy, immunotherapy or investigational drug concurrent or within 28 days or 5 half-lives of the drug (whichever is shorter) before the first study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) (Parts 1 and 2) | Up to 36 months
Percentage of Participants with Dose-Limiting Toxicities (DLTs) (Parts 1 and 2) | Up to 36 months
Objective Response Rate (ORR) (Part 3) | Up to 48 months

SECONDARY OUTCOMES:
Area Under The Curve (AUC) of RO7300490 (Parts 1, 2 and 3) | Up to 48 months
Minimum Concentration (Cmin) of RO7300490 (Parts 1, 2 and 3) | Up to 48 months
Maximum Concentration (Cmax) of RO7300490 (Parts 1, 2 and 3) | Up to 48 months
Clearance (CL) of RO7300490 (Parts 1, 2 and 3) | Up to 48 months
Volume of Distribution at Steady State (Vss) of RO7300490 (Parts 1, 2 and 3) | Up to 48 months
Percentage of Participants with Anti-RO7300490 Antibodies (Parts 1, 2 and 3) | Up to 48 months
Objective Response Rate (ORR) (Parts 1 and 2) | Up to 48 months
Disease Control Rate (DCR) (Parts 1, 2 and 3) | Up to 48 months
Duration of Response (DOR) (Parts 1, 2 and 3) | Up to 48 months
Progression-Free Survival (PFS) On-Treatment (Parts 1, 2 and 3) | Up to 48 months
Percentage of Participants With Adverse Events (AEs) (Part 3) | Up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Rigshospitalet; Fase 1 Enhed - Onkologi, København Ø, Denmark
- Gustave Roussy, Villejuif, France
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Clinica Universidad de Navarra Madrid; Servicio de Oncología, Madrid
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
- United Kingdom (3):
  - Western General Hospital; Edinburgh Cancer Center, Edinburgh
  - Guys and St Thomas Hospital; OHCT Clinical Trials, London
  - Christie Hospital NHS Trust; Experimental Cancer Medicine Team, Manchester